CLINICAL TRIAL: NCT00539461
Title: Sifrol® (Pramipexole) Impact on RLS Related Quality of Life: A 12-weeks Observational Study in Patients With Primary RLS
Brief Title: Non-interventional Observational Study of Pramipexole in Restless Legs Syndrome: Impact on Quality of Life
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.638
Record Dates: First submitted 2007-09-28; First posted 2007-10-04 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
In this German non-interventional observational study 1980 patients diagnosed with Restless Legs Syndrome (RLS) will be investigated by 990 General Practitioners across all federal states in Germany. Both moderate to severe RLS patients, with or without previous RLS treatment, suffering from RLS symptoms like a desire to move the extremities usually associated with some discomfort, motor restlessness and worsening of symptoms at rest with at least temporary relief by activity, worsening of symptoms later in the day or at night, are eligible for this study, if it is planned to initiate therapy with pramipexole or to add pramipexole to a previously given, insufficient therapy. Three visits are planned to be documented in this PMS study, one baseline visit, visit two after the end of pramipexole titration and visit three after 12 weeks of treatment. Evaluations and visits are to be carried out and documented only if part of routine medical practice. The main goal of observational studies is to determine how pramipexole treatment works when applied in actual practice and thus maximise external validity. In actual practice patients who have been excluded in the clinical registration trials of PPX in moderate to severe primary RLS (i.e. those with certain disease histories, co-morbidities and/or demographic characteristics) will be treated with PPX. Thus in addition during this observational study information on the efficacy and safety of PPX in those patients will be obtained. The objectives of this PMS study are:

* To evaluate the treatment effect of pramipexole on RLS severity and general improvement as measured by IRLS and CGI-I.
* To evaluate quality of life of RLS patients as measured by the Restless Legs Syndrome Quality of Life questionnaire (RLS-QoL).
* To evaluate the safety profile of PPX in a natural study population.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of primary RLS
2. Indication for RLS treatment with Sifrol® (pramipexole)
3. Male or female patients aged at least 18 years.

Exclusion Criteria:

1. Any contraindications according to the Summary of Product Characteristics (SPC): hypersensitivity to pramipexole or to any of the excipients.
2. Ongoing treatment with Sifrol® (pramipexole).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RLS patients
Sampling Method: Non-Probability Sample
Enrollment: 2023 (Actual)
Dates: Start 2007-02; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IRLS total score after 12 weeks | 12 weeks
CGI-I responder rate after 12 weeks | 12 weeks
Time to reach maintenance dose | 12 weeks
Change from baseline in RLS-QoL total score after 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in IRLS score after 1-4 weeks | 4 weeks
Change in IRLS items after 12 weeks | 12 weeks
Final dose distribution | 12 weeks
Incidence, relationship and seriousness of adverse events | 12 weeks
Number of premature discontinuations | 12 weeks

CONTACTS AND LOCATIONS:
Locations (317):
- Germany (317):
  - Boehringer Ingelheim Investigational Site, Aalen
  - Boehringer Ingelheim Investigational Site, Aarbergen
  - Boehringer Ingelheim Investigational Site, Adendorf
  - Boehringer Ingelheim Investigational Site, Aham
  - Boehringer Ingelheim Investigational Site, Ahaus
  - Boehringer Ingelheim Investigational Site, Ahlen
  - Boehringer Ingelheim Investigational Site, Ahorntal
  - Boehringer Ingelheim Investigational Site, Aichach
  - Boehringer Ingelheim Investigational Site, Aislingen
  - Boehringer Ingelheim Investigational Site, Albstadt
  - Boehringer Ingelheim Investigational Site, Aldenhoven
  - Boehringer Ingelheim Investigational Site, Aldingen
  - Boehringer Ingelheim Investigational Site, Alfeld
  - Boehringer Ingelheim Investigational Site, Alpirsbach
  - Boehringer Ingelheim Investigational Site, Alsdorf
  - Boehringer Ingelheim Investigational Site, Altena
  - Boehringer Ingelheim Investigational Site, Altenstadt
  - Boehringer Ingelheim Investigational Site, Altomünster
  - Boehringer Ingelheim Investigational Site, Alveslohe
  - Boehringer Ingelheim Investigational Site, Amberg
  - Boehringer Ingelheim Investigational Site, Ammerbuch
  - Boehringer Ingelheim Investigational Site, Andernach
  - Boehringer Ingelheim Investigational Site, Anklam
  - Boehringer Ingelheim Investigational Site, Apolda
  - Boehringer Ingelheim Investigational Site, Armsheim
  - Boehringer Ingelheim Investigational Site, Arzberg
  - Boehringer Ingelheim Investigational Site, Aschaffenburg
  - Boehringer Ingelheim Investigational Site, Aschersleben
  - Boehringer Ingelheim Investigational Site, Aschheim
  - Boehringer Ingelheim Investigational Site, Attendorn
  - Boehringer Ingelheim Investigational Site, Auerbach
  - Boehringer Ingelheim Investigational Site, Augsburg
  - Boehringer Ingelheim Investigational Site, Aurich
  - Boehringer Ingelheim Investigational Site, Babensham
  - Boehringer Ingelheim Investigational Site, Backnang
  - Boehringer Ingelheim Investigational Site, Bad Arolsen
  - Boehringer Ingelheim Investigational Site, Bad Berleburg
  - Boehringer Ingelheim Investigational Site, Bad Bevensen
  - Boehringer Ingelheim Investigational Site, Bad Düben
  - Boehringer Ingelheim Investigational Site, Bad Dürrenberg
  - Boehringer Ingelheim Investigational Site, Bad Dürrheim
  - Boehringer Ingelheim Investigational Site, Bad Ems
  - Boehringer Ingelheim Investigational Site, Bad Essen
  - Boehringer Ingelheim Investigational Site, Bad Kreuznach
  - Boehringer Ingelheim Investigational Site, Bad Laasphe
  - Boehringer Ingelheim Investigational Site, Bad Langensalza
  - Boehringer Ingelheim Investigational Site, Bad Lausick
  - Boehringer Ingelheim Investigational Site, Bad Münstereifel
  - Boehringer Ingelheim Investigational Site, Bad Oeynhausen
  - Boehringer Ingelheim Investigational Site, Bad Salzungen
  - Boehringer Ingelheim Investigational Site, Bad Schwalbach
  - Boehringer Ingelheim Investigational Site, Bad Schwartau
  - Boehringer Ingelheim Investigational Site, Bad Segeberg
  - Boehringer Ingelheim Investigational Site, Bad Tennstedt
  - Boehringer Ingelheim Investigational Site, Bad Waldsee
  - Boehringer Ingelheim Investigational Site, Baden-Baden
  - Boehringer Ingelheim Investigational Site, Bahrdorf
  - Boehringer Ingelheim Investigational Site, Baltmannsweiler
  - Boehringer Ingelheim Investigational Site, Bamberg
  - Boehringer Ingelheim Investigational Site, Barleben
  - Boehringer Ingelheim Investigational Site, Baunatal
  - Boehringer Ingelheim Investigational Site, Bautzen
  - Boehringer Ingelheim Investigational Site, Bayreuth
  - Boehringer Ingelheim Investigational Site, Bärnau
  - Boehringer Ingelheim Investigational Site, Beckum
  - Boehringer Ingelheim Investigational Site, Beeskow
  - Boehringer Ingelheim Investigational Site, Bellheim
  - Boehringer Ingelheim Investigational Site, Belm
  - Boehringer Ingelheim Investigational Site, Bensheim
  - Boehringer Ingelheim Investigational Site, Berching
  - Boehringer Ingelheim Investigational Site, Bergfelde
  - Boehringer Ingelheim Investigational Site, Bergheim
  - Boehringer Ingelheim Investigational Site, Bergisch Gladbach
  - Boehringer Ingelheim Investigational Site, Berkheim
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Berne
  - Boehringer Ingelheim Investigational Site, Bernsdorf
  - Boehringer Ingelheim Investigational Site, Betzdorf
  - Boehringer Ingelheim Investigational Site, Biebertal
  - Boehringer Ingelheim Investigational Site, Bielefeld
  - Boehringer Ingelheim Investigational Site, Bienenbüttel
  - Boehringer Ingelheim Investigational Site, Bippen
  - Boehringer Ingelheim Investigational Site, Birkenfeld
  - Boehringer Ingelheim Investigational Site, Birkenwerder
  - Boehringer Ingelheim Investigational Site, Blankenhain
  - Boehringer Ingelheim Investigational Site, Blaustein
  - Boehringer Ingelheim Investigational Site, Blieskastel
  - Boehringer Ingelheim Investigational Site, Bobritzsch
  - Boehringer Ingelheim Investigational Site, Bocholt
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site, Bockenem
  - Boehringer Ingelheim Investigational Site, Bodelshausen
  - Boehringer Ingelheim Investigational Site, Bodenfelde
  - Boehringer Ingelheim Investigational Site, Bodenkirchen
  - Boehringer Ingelheim Investigational Site, Bodenwöhr
  - Boehringer Ingelheim Investigational Site, Bodman-Ludwigshafen
  - Boehringer Ingelheim Investigational Site, Bollendorf
  - Boehringer Ingelheim Investigational Site, Bonn
  - Boehringer Ingelheim Investigational Site, Bopfingen
  - Boehringer Ingelheim Investigational Site, Borgholzhausen
  - Boehringer Ingelheim Investigational Site, Borken
  - Boehringer Ingelheim Investigational Site, Borna
  - Boehringer Ingelheim Investigational Site, Bornheim
  - Boehringer Ingelheim Investigational Site, Bottendorf
  - Boehringer Ingelheim Investigational Site, Bottmersdorf
  - Boehringer Ingelheim Investigational Site, Bottrop
  - Boehringer Ingelheim Investigational Site, Bovenden
  - Boehringer Ingelheim Investigational Site, Böhlen
  - Boehringer Ingelheim Investigational Site, Bösel
  - Boehringer Ingelheim Investigational Site, Brake
  - Boehringer Ingelheim Investigational Site, Brandenburg
  - Boehringer Ingelheim Investigational Site, Brannenburg
  - Boehringer Ingelheim Investigational Site, Braunschweig
  - Boehringer Ingelheim Investigational Site, Brechen
  - Boehringer Ingelheim Investigational Site, Breitenbrunn
  - Boehringer Ingelheim Investigational Site, Bremen
  - Boehringer Ingelheim Investigational Site, Bremerhaven
  - Boehringer Ingelheim Investigational Site, Brensbach
  - Boehringer Ingelheim Investigational Site, Breuberg
  - Boehringer Ingelheim Investigational Site, Bruchköbel
  - Boehringer Ingelheim Investigational Site, Brunsbüttel
  - Boehringer Ingelheim Investigational Site, Buchbach
  - Boehringer Ingelheim Investigational Site, Buckow
  - Boehringer Ingelheim Investigational Site, Buedelsdorf
  - Boehringer Ingelheim Investigational Site, Burg
  - Boehringer Ingelheim Investigational Site, Burgau
  - Boehringer Ingelheim Investigational Site, Burgdorf, Hanover
  - Boehringer Ingelheim Investigational Site, Burgpreppach
  - Boehringer Ingelheim Investigational Site, Burtenbach
  - Boehringer Ingelheim Investigational Site, Buttstädt
  - Boehringer Ingelheim Investigational Site, Butzbach
  - Boehringer Ingelheim Investigational Site, Bückeburg
  - Boehringer Ingelheim Investigational Site, Bünde
  - Boehringer Ingelheim Investigational Site, Büttelborn
  - Boehringer Ingelheim Investigational Site, Cadolzburg
  - Boehringer Ingelheim Investigational Site, Calbe
  - Boehringer Ingelheim Investigational Site, Calberlah
  - Boehringer Ingelheim Investigational Site, Castrop-Rauxel
  - Boehringer Ingelheim Investigational Site, Celle
  - Boehringer Ingelheim Investigational Site, Chemnitz
  - Boehringer Ingelheim Investigational Site, Cochem
  - Boehringer Ingelheim Investigational Site, Coppenbrügge
  - Boehringer Ingelheim Investigational Site, Crimmitschau
  - Boehringer Ingelheim Investigational Site, Crivitz
  - Boehringer Ingelheim Investigational Site, Cuxhaven
  - Boehringer Ingelheim Investigational Site, Dabel
  - Boehringer Ingelheim Investigational Site, Darmstadt
  - Boehringer Ingelheim Investigational Site, Dassow
  - Boehringer Ingelheim Investigational Site, Datteln
  - Boehringer Ingelheim Investigational Site, Daun
  - Boehringer Ingelheim Investigational Site, Deggendorf
  - Boehringer Ingelheim Investigational Site, Deidesheim
  - Boehringer Ingelheim Investigational Site, Deining
  - Boehringer Ingelheim Investigational Site, Delitzsch
  - Boehringer Ingelheim Investigational Site, Demen
  - Boehringer Ingelheim Investigational Site, Denkendorf
  - Boehringer Ingelheim Investigational Site, Dessau
  - Boehringer Ingelheim Investigational Site, Detmold
  - Boehringer Ingelheim Investigational Site, Dettenheim
  - Boehringer Ingelheim Investigational Site, Deuben
  - Boehringer Ingelheim Investigational Site, Deutzen
  - Boehringer Ingelheim Investigational Site, Diepholz
  - Boehringer Ingelheim Investigational Site, Dillingen
  - Boehringer Ingelheim Investigational Site, Dingolfing
  - Boehringer Ingelheim Investigational Site, Dinkelsbühl
  - Boehringer Ingelheim Investigational Site, Dinslaken
  - Boehringer Ingelheim Investigational Site, Dissen
  - Boehringer Ingelheim Investigational Site, Dogern
  - Boehringer Ingelheim Investigational Site, Dollern
  - Boehringer Ingelheim Investigational Site, Donaueschingen
  - Boehringer Ingelheim Investigational Site, Dormagen
  - Boehringer Ingelheim Investigational Site, Dornstetten
  - Boehringer Ingelheim Investigational Site, Dorsten
  - Boehringer Ingelheim Investigational Site, Dortmund
  - Boehringer Ingelheim Investigational Site, Dörentrup
  - Boehringer Ingelheim Investigational Site, Dörpen
  - Boehringer Ingelheim Investigational Site, Dreieich
  - Boehringer Ingelheim Investigational Site, Drensteinfurt
  - Boehringer Ingelheim Investigational Site, Dresden
  - Boehringer Ingelheim Investigational Site, Driedorf
  - Boehringer Ingelheim Investigational Site, Duderstadt
  - Boehringer Ingelheim Investigational Site, Duisburg
  - Boehringer Ingelheim Investigational Site, Dummerstorf
  - Boehringer Ingelheim Investigational Site, Düren
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Boehringer Ingelheim Investigational Site, Ebergötzen
  - Boehringer Ingelheim Investigational Site, Ebermannstadt
  - Boehringer Ingelheim Investigational Site, Eberstadt
  - Boehringer Ingelheim Investigational Site, Ebhausen
  - Boehringer Ingelheim Investigational Site, Edewecht
  - Boehringer Ingelheim Investigational Site, Edling
  - Boehringer Ingelheim Investigational Site, Egelsbach
  - Boehringer Ingelheim Investigational Site, Ehingen
  - Boehringer Ingelheim Investigational Site, Eilenburg
  - Boehringer Ingelheim Investigational Site, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site, Eiterfeld
  - Boehringer Ingelheim Investigational Site, Eitorf
  - Boehringer Ingelheim Investigational Site, Ellwangen
  - Boehringer Ingelheim Investigational Site, Elmshorn
  - Boehringer Ingelheim Investigational Site, Emersacker
  - Boehringer Ingelheim Investigational Site, Emmendingen
  - Boehringer Ingelheim Investigational Site, Emsdetten
  - Boehringer Ingelheim Investigational Site, Enger
  - Boehringer Ingelheim Investigational Site, Enkenbach-Alsenborn
  - Boehringer Ingelheim Investigational Site, Ennepetal
  - Boehringer Ingelheim Investigational Site, Ennigerloh
  - Boehringer Ingelheim Investigational Site, Eppstein
  - Boehringer Ingelheim Investigational Site, Erding
  - Boehringer Ingelheim Investigational Site, Erftstadt
  - Boehringer Ingelheim Investigational Site, Erkrath
  - Boehringer Ingelheim Investigational Site, Erligheim
  - Boehringer Ingelheim Investigational Site, Erndtebrück
  - Boehringer Ingelheim Investigational Site, Erolzheim
  - Boehringer Ingelheim Investigational Site, Eschborn
  - Boehringer Ingelheim Investigational Site, Eschelbronn
  - Boehringer Ingelheim Investigational Site, Eschweiler
  - Boehringer Ingelheim Investigational Site, Eslohe
  - Boehringer Ingelheim Investigational Site, Espenhain
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Euskirchen
  - Boehringer Ingelheim Investigational Site, Filderstadt
  - Boehringer Ingelheim Investigational Site, Floh-Seligenthal
  - Boehringer Ingelheim Investigational Site, Flöha
  - Boehringer Ingelheim Investigational Site, Forbach
  - Boehringer Ingelheim Investigational Site, Forchheim
  - Boehringer Ingelheim Investigational Site, Frankenberg
  - Boehringer Ingelheim Investigational Site, Frankenthal
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Freiberg
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site, Freigericht
  - Boehringer Ingelheim Investigational Site, Freudenstadt
  - Boehringer Ingelheim Investigational Site, Freyung
  - Boehringer Ingelheim Investigational Site, Friedland
  - Boehringer Ingelheim Investigational Site, Friedrichshafen
  - Boehringer Ingelheim Investigational Site, Friedrichsthal
  - Boehringer Ingelheim Investigational Site, Frohburg
  - Boehringer Ingelheim Investigational Site, Fulda
  - Boehringer Ingelheim Investigational Site, Furtwangen im Schwarzwald
  - Boehringer Ingelheim Investigational Site, Fürstenwalde
  - Boehringer Ingelheim Investigational Site, Füssen
  - Boehringer Ingelheim Investigational Site, Gangelt
  - Boehringer Ingelheim Investigational Site, Gardelegen
  - Boehringer Ingelheim Investigational Site, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site, Gars
  - Boehringer Ingelheim Investigational Site, Gebesee
  - Boehringer Ingelheim Investigational Site, Geesthacht
  - Boehringer Ingelheim Investigational Site, Gelbensande
  - Boehringer Ingelheim Investigational Site, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site, Gensingen
  - Boehringer Ingelheim Investigational Site, Georgsmarienhütte
  - Boehringer Ingelheim Investigational Site, Gera
  - Boehringer Ingelheim Investigational Site, Gerbstedt
  - Boehringer Ingelheim Investigational Site, Germering
  - Boehringer Ingelheim Investigational Site, Germersheim
  - Boehringer Ingelheim Investigational Site, Gevelsberg
  - Boehringer Ingelheim Investigational Site, Giessen
  - Boehringer Ingelheim Investigational Site, Gifhorn
  - Boehringer Ingelheim Investigational Site, Gilserberg
  - Boehringer Ingelheim Investigational Site, Gladbeck
  - Boehringer Ingelheim Investigational Site, Gleichen
  - Boehringer Ingelheim Investigational Site, Goch
  - Boehringer Ingelheim Investigational Site, Gochsheim
  - Boehringer Ingelheim Investigational Site, Gomaringen
  - Boehringer Ingelheim Investigational Site, Göllheim
  - Boehringer Ingelheim Investigational Site, Göllingen
  - Boehringer Ingelheim Investigational Site, Göttingen
  - Boehringer Ingelheim Investigational Site, Grafenau
  - Boehringer Ingelheim Investigational Site, Gransee
  - Boehringer Ingelheim Investigational Site, Grassau
  - Boehringer Ingelheim Investigational Site, Greiz
  - Boehringer Ingelheim Investigational Site, Greven
  - Boehringer Ingelheim Investigational Site, Grevesmühlen
  - Boehringer Ingelheim Investigational Site, Griesheim
  - Boehringer Ingelheim Investigational Site, Gronau
  - Boehringer Ingelheim Investigational Site, Groß Grönau
  - Boehringer Ingelheim Investigational Site, Groß Quenstedt
  - Boehringer Ingelheim Investigational Site, Groß-Zimmern
  - Boehringer Ingelheim Investigational Site, Großalmerode
  - Boehringer Ingelheim Investigational Site, Großbottwar
  - Boehringer Ingelheim Investigational Site, Großefehn
  - Boehringer Ingelheim Investigational Site, Großhabersdorf
  - Boehringer Ingelheim Investigational Site, Großkorbetha
  - Boehringer Ingelheim Investigational Site, Großlangheim
  - Boehringer Ingelheim Investigational Site, Grömitz
  - Boehringer Ingelheim Investigational Site, Grünbach
  - Boehringer Ingelheim Investigational Site, Gummersbach
  - Boehringer Ingelheim Investigational Site, Güstrow
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Hagen
  - Boehringer Ingelheim Investigational Site, Haigerloch
  - Boehringer Ingelheim Investigational Site, Haldensleben I
  - Boehringer Ingelheim Investigational Site, Halle
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hamm
  - Boehringer Ingelheim Investigational Site, Hamminkeln
  - Boehringer Ingelheim Investigational Site, Hanau
  - Boehringer Ingelheim Investigational Site, Hanerau-Hademarschen
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Harpstedt
  - Boehringer Ingelheim Investigational Site, Harsefeld
  - Boehringer Ingelheim Investigational Site, Harsewinkel
  - Boehringer Ingelheim Investigational Site, Haselünne
  - Boehringer Ingelheim Investigational Site, Hattersheim
  - Boehringer Ingelheim Investigational Site, Hattingen
  - Boehringer Ingelheim Investigational Site, Havixbeck
  - Boehringer Ingelheim Investigational Site, Hedersleben
  - Boehringer Ingelheim Investigational Site, Heek
  - Boehringer Ingelheim Investigational Site, Heide
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Heilbronn
  - Boehringer Ingelheim Investigational Site, Heimsheim
  - Boehringer Ingelheim Investigational Site, Heinsberg
  - Boehringer Ingelheim Investigational Site, Hellenthal
  - Boehringer Ingelheim Investigational Site, Hermaringen
  - Boehringer Ingelheim Investigational Site, Huska